CLINICAL TRIAL: NCT01556971
Title: A Controlled Study of the Efficacy of Botulinum Toxin A (Botox) for the Treatment of Major Depressive Disorder (MDD)
Brief Title: Efficacy Study of Botox for Depression
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Capital Clinical Research Associates, LLC (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: Botox 5515
Record Dates: First submitted 2012-03-15; First posted 2012-03-19 (Estimated); Last update posted 2012-03-19 (Estimated); Status verified 2012-03

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Botox (Active Comparator): The study will be divided randomly into two groups of equal number; one arm will receive a Botox injection; the other will receive saline solution injection
  Interventions: Drug: Botox
- Saline Solution (Placebo Comparator): A saline solution will be injected in to the procerus and corrugator supercilii frown muscles of randomly chosen study participants.
  Interventions: Drug: Saline Solution

INTERVENTIONS:
Drug: Botox — Appropriate patients will randomly receive 29 units of Botox or a saline solution injected in to the procerus and corrugator supercilii frown muscles.
  Arms: Botox
Drug: Saline Solution — 29 units of saline solution will be injected in to the procerus and corrugator supercilii frown muscles of randomly chosen study participants.
  Arms: Saline Solution

SUMMARY:
The objective of this proposed study is to obtain data on the efficacy of Botox in reducing symptoms of MDD in male and female patients between the ages of 18 and 65 years old.

The secondary object is to visually assess each patient's frown before and after the Botox injection to determine if there is a correlation between changes in the frown and changes in mood. The patients will be photographed at screening, visit 2 and 3. Their frown lines will be compared to determine if there is a visible improvement in the frown lines corresponding to an improvement in the efficacy rating scores.

DETAILED DESCRIPTION:
This will be a double-blind study. To maintain the blinding of the study, none of the investigators who are assessing depression scores will be aware of the injection status of the patients. In addition, to maintain patient blinding, the patients will not be educated as to possible expected outcomes on facial expressions. Unless specifically informed, patients are generally unaware of the facial movement that is inhibited by Botulinum Toxin A. An unblinded physician will act as pharmacist for the study preparing the active drug and the placebo for the injections.

Duration of Treatment: The study will be divided into three phases: screening and enrollment, treatment and follow-up. Patients who meet all criteria will be randomized at the screening visit. The treatment phase will last six (6) weeks after the investigational product is administered during which the patients will return to for a visit at week 3. Subjects will return to the office for a discontinuation visit at week six.

General Design and Methodology: At screening, patients will sign consent and be diagnosed by means of the M.I.N.I. They will be assessed by a clinician who will perform the MADRS and CGI-S which are standardized ratings. They will complete the patient-rated BDI. Subjects will provide a urine sample for drug screening. WOCBP will be given a pregnancy test. Patients who meet all criteria will be randomly assigned to receive either the investigational product or placebo. The study medication or placebo will be injected into the procerus and corrugator supercilii frown muscles of each patient by a physician or physician's assistant. Each patient face will be photographed at this an all visits. Three weeks ± 7 days following the injection, each patient will return to the office where a clinician will administer the MADRS and the CGI-I. The patient will complete the BDI and adverse events (AEs) and concomitant medications will be collected.

Six weeks ± 7 days following the injection, patients will return to the office where the clinician will administer the MADRS and CGI-I, collect AEs and concomitant medications. The patients will complete the BDI. All patients, whether on the active drug or the placebo, will be given a voucher which they may use for a free Botox injection at week 8, if , in the judgment of the investigator, it will be beneficial to the patient.

Diagnosis and Criteria for Inclusion: Patients will be included in this study if they meet all of the following criteria:

* Written informed consent is obtained;
* They are a 18 to 65 years old;
* They meet DSM-IV criteria for MDD as diagnosed by the MINI at screening, and, their current episode must be at least one month in length;
* They have a MADRS score of ≥ 26 at screening;
* They have ≥ 4 on the CGI-S at screening
* Women of childbearing potential (WOCBP) are on an acceptable form of birth control and are not pregnant or lactating;
* They are judged by the investigator to have the capacity to understand the nature of the study;
* They are willing to comply with all the requirements of the study.
* They are considered by the investigator to be likely to adhere to the protocol.

Criteria for Exclusion: Patients will be excluded from this study if they meet any of the following criteria:

* They have been treated with botulinum toxin A in the 12 months prior to screening;
* They have another Axis I disorder as a principal diagnosis in the 6 months prior to screening;
* They have a history of substance abuse or dependency in the 2 months prior to screening (recreational use of illicit drugs may be permissible, at the discretion of the investigator);
* They test positive for illicit drugs on urine drug screen, and this has not been adequately explained to the satisfaction of the investigator;
* They endorse MADRS item 10 (suicidal ideas) at a level of 5 or more or have attempted suicide in the six months prior to screening;
* They are considered to be at a significant risk of committing homicide;
* They have an unstable medical condition;
* Women of childbearing potential (WOCBP) who are pregnant or are considering becoming pregnant during the length of the study;
* They are regarded, for any reason by the principal investigator as being an unsuitable candidate for the protocol.
* There has been a change in their medication or psychotherapy treatment regimen in the month preceding screening;
* They have proved to be refractory to three or more adequate antidepressant treatments with methods that have different mechanisms of action.

ELIGIBILITY:
Inclusion Criteria:• Written informed consent is obtained;

* They are a 18 to 65 years old;
* They meet DSM-IV criteria for MDD as diagnosed by the MINI at screening, and, their current episode must be at least one month in length;
* They have a MADRS score of ≥ 26 at screening;
* They have ≥ 4 on the CGI-S at screening
* Women of childbearing potential (WOCBP) are on an acceptable form of birth control and are not pregnant or lactating;
* They are judged by the investigator to have the capacity to understand the nature of the study;
* They are willing to comply with all the requirements of the study.
* They are considered by the investigator to be likely to adhere to the protocol.

Exclusion Criteria:• They have been treated with botulinum toxin A in the 12 months prior to screening;

* They have another Axis I disorder as a principal diagnosis in the 6 months prior to screening;
* They have a history of substance abuse or dependency in the 2 months prior to screening (recreational use of illicit drugs may be permissible, at the discretion of the investigator);
* They test positive for illicit drugs on urine drug screen, and this has not been adequately explained to the satisfaction of the investigator;
* They endorse MADRS item 10 (suicidal ideas) at a level of 5 or more or have attempted suicide in the six months prior to screening;
* They are considered to be at a significant risk of committing homicide;
* They have an unstable medical condition;
* Women of childbearing potential (WOCBP) who are pregnant or are considering becoming pregnant during the length of the study;
* They are regarded, for any reason by the principal investigator as being an unsuitable candidate for the protocol.
* There has been a change in their medication or psychotherapy treatment regimen in the month preceding screening;
* They have proved to be refractory to three or more adequate antidepressant treatments with methods that have different mechanisms of action.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-06 (Estimated); Study Completion 2012-06 (Estimated)

PRIMARY OUTCOMES:
MADRS | Patients will be followed for up to 10 weeks
  Efficacy will be assessed using: the Montgomery-Asberg Depression Rating Scale (MADRS) screening, visit 2 and discontinuation
Beck Depression Inventory | Patients will be followed for up to 10 weeks
  Efficacy will be assessed using the patient-rated Beck Depression Inventory II (BDI) at screening, visit 2 and discontinuation.
CGI-I | Patients will be followed for up to 10 weeks
  Efficacy will be assessed using the Clinical Global Impression-Improvement (CGI-I) at visit 2 and discontinuation

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Z Rosenthal, MD, Principal Investigator — Capital Clinical Research Association
Locations (2):
- United States (2):
  - Chevy Chase Cosmetic Center, Chevy Chase, Maryland
  - Capital Clinical Research Associates, LLC, Rockville, Maryland

REFERENCES:
- [Derived] Finzi E, Rosenthal NE. Treatment of depression with onabotulinumtoxinA: a randomized, double-blind, placebo controlled trial. J Psychiatr Res. 2014 May;52:1-6. doi: 10.1016/j.jpsychires.2013.11.006. Epub 2013 Dec 1. PMID 24345483